CLINICAL TRIAL: NCT03110770
Title: VRC 705: A Phase 2/2B, Randomized Trial to Evaluate the Safety, Immunogenicity and Efficacy of a Zika Virus DNA Vaccine in Healthy Adults and Adolescents
Brief Title: VRC 705: A Zika Virus DNA Vaccine in Healthy Adults and Adolescents
Acronym: DNA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Prevention
Other Study IDs: VRC 705
Record Dates: First submitted 2017-03-28; First posted 2017-04-12 (Actual); Results first posted 2020-12-04 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Zika Virus; Zika Virus Infection; Virus Diseases; Flavivirus Infections; Flaviviral Diseases; Flaviviridae Infections; RNA Virus Infections
Keywords: Flavivirus; Zika; Vaccine; Physiological Effects of Drugs; Immunologic Factors; Virus-like Particles; Zika vaccine
MeSH Terms: conditions — Zika Virus Infection; Virus Diseases; Flavivirus Infections; Flaviviridae Infections; RNA Virus Infections

STUDY DESIGN:
Intervention Model Description: Part A participants (n=90) were randomized to study groups at a 1:1:1 ratio to receive a 4 mg or 8 mg dose of vaccine split between 2 or 4 injections. In Part B, participants (n=2338) were randomized to vaccine or placebo in a 1:1 ratio to receive a 4 mg (1 mL) dose of vaccine or 1 mL of placebo split between 2 injections. The vaccine dose and number of injections in Part B was determined by preliminary data from the Phase 1 trial and from Part A.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Part A was open-label. For Part A, the participant, investigator and outcome assessor knew what the participant received.
  Part B injections were prepared by an unblinded site pharmacist or designee who was not involved in any participant assessments and did not discuss randomizations with study clinicians. Participants, study personnel, site data entry personnel, and laboratory personnel performing immunologic assays were blinded to the treatment assignment of all product administrations. The investigational new drug (IND) Sponsor unblinded treatment assignments for Part B at the end of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part A, Group 1: VRC-ZKADNA090-00-VP (4 mg), 2 injections (Experimental): Zika virus wildtype (ZIKVwt) DNA vaccine (VRC-ZKADNA090-00-VP), in 2 limbs (both arms) on Day 0, Day 28 (+/-7 days), and Day 56 (-7/+14 days); 4 mg of vaccine administered intramuscularly (IM) by a needle-free injection device
  Interventions: Biological: VRC-ZKADNA090-00-VP
- Part A, Group 2: VRC-ZKADNA090-00-VP (4 mg), 4 injections (Experimental): ZIKVwt DNA vaccine (VRC-ZKADNA090-00-VP), in 4 limbs (both arms and legs) on Day 0, Day 28 (+/-7 days), and Day 56 (-7/+14 days); 4 mg of vaccine administered IM by a needle-free injection device
  Interventions: Biological: VRC-ZKADNA090-00-VP
- Part A, Group 3: VRC-ZKADNA090-00-VP (8 mg), 4 injections (Experimental): ZIKVwt DNA vaccine (VRC-ZKADNA090-00-VP), in 4 limbs (both arms and legs) on Day 0, Day 28 (+/-7 days), and Day 56 (-7/+14 days); 8 mg of vaccine administered IM by a needle-free injection device
  Interventions: Biological: VRC-ZKADNA090-00-VP
- Part B, Group 4: VRC-ZKADNA090-00-VP (4 mg), 2 injections (Experimental): ZIKVwt DNA vaccine (VRC-ZKADNA090-00-VP), in 2 limbs (both arms) on Day 0, Day 28 (+/-7 days), and Day 56 (-7/+14 days); 4 mg of vaccine administered IM by a needle-free injection device
  Interventions: Biological: VRC-ZKADNA090-00-VP
- Part B, Group 5: Placebo (VRC-PBSPLA043-00-VP), 2 injections (Placebo Comparator): Sterile phosphate-buffered saline (PBS) (VRC-PBSPLA043-00-VP), the placebo, in 2 limbs (both arms) on Day 0, Day 28 (+/-7 days), and Day 56 (-7/+14 days); 1 mL of placebo administered IM by a needle-free injection device
  Interventions: Other: VRC-PBSPLA043-00-VP

INTERVENTIONS:
Biological: VRC-ZKADNA090-00-VP — VRC-ZKADNA090-00-VP is composed of a single closed-circular DNA plasmid (VRC 5283) that encodes with wild type (wt) precursor transmembrane M (prM) and envelope (E) proteins from the H/PF/2013 strain of ZIKV
  Arms: Part A, Group 1: VRC-ZKADNA090-00-VP (4 mg), 2 injections; Part A, Group 2: VRC-ZKADNA090-00-VP (4 mg), 4 injections; Part A, Group 3: VRC-ZKADNA090-00-VP (8 mg), 4 injections; Part B, Group 4: VRC-ZKADNA090-00-VP (4 mg), 2 injections
Other: VRC-PBSPLA043-00-VP — A sterile phosphate-buffered saline (PBS) prepared for human administration as a placebo
  Other Names: Placebo
  Arms: Part B, Group 5: Placebo (VRC-PBSPLA043-00-VP), 2 injections

SUMMARY:
This was a multicenter, randomized study to evaluate the safety, immunogenicity, and efficacy of VRC-ZKADNA090-00-VP (Zika virus wildtype DNA vaccine) or placebo. In Part A, the primary objective was to evaluate the safety and tolerability of the vaccine in different vaccination regimens. In Part B, the primary objectives were to evaluate the safety and efficacy of the vaccine compared to placebo.

DETAILED DESCRIPTION:
This was a multicenter, randomized study to evaluate safety, immunogenicity, and efficacy of a 3-dose vaccination regimen with the Zika virus wildtype (ZIKVwt) DNA vaccine (VRC-ZKADNA090-00-VP) or placebo (VRC-PBSPLA043-00-VP). The placebo was a sterile phosphate-buffered saline (PBS). The hypotheses were that the ZIKVwt DNA vaccine would be safe and would elicit a ZIKV-specific immune response.

Participants received study product intramuscularly (IM) in the limbs as specified by the group assignment by PharmaJet needle-free device. In Part A, 90 participants were randomized to vaccine at a 1:1:1 ratio to receive a 4 mg dose split between 2 injections, 4 mg dose split between 4 injections or 8 mg dose split between 4 injections. In Part B, 2338 participants were randomized to vaccine or placebo in a 1:1 ratio to receive a 4 mg (1 mL) dose of vaccine or 1 mL of placebo split between 2 injections. The vaccine dose and administration plan for Part B was selected based on Part A and Phase 1 data.

Vaccine safety and tolerability were assessed by monitoring of clinical and laboratory parameters throughout the study. Solicited reactogenicity symptoms were collected for 7 days after each product administration. The study schedule included clinic visits with safety and immunogenicity blood samples collected at particular time points.

Vaccine efficacy was evaluated in Part B by comparing incidence of virologic ZIKV cases between vaccine and placebo groups. During the study, when participants exhibited any possible symptom of ZIKV infection, they were evaluated by blood and urine ZIKV polymerase chain reaction (PCR). Stored blood samples were also assessed retrospectively by ZIKV PCR to identify possible asymptomatic cases. A Data and Safety Monitoring Board (DSMB) oversaw the study.

ELIGIBILITY:
Inclusion Criteria:

A participant must meet all of the following criteria:

Part A:

* 18 to 35 years of age
* Available for clinical follow-up through Study Week 32
* Accessible injection sites on each limb as follows: 1 injection site in the deltoid muscle of each arm and 1 injection site in the vastus lateralis muscle of each anterolateral thigh

Part B:

* 15 to 35 years of age
* Available for clinical follow-up through Study Week 96
* Accessible injection sites on the deltoid muscle of each arm. Injection in the vastus lateralis muscle of the anterolateral thighs may have been allowed with IND Sponsor approval if an injection site on each deltoid muscle was not available.

Part A and B:

* Able to provide proof of identity to the satisfaction of the clinician completing the enrollment process
* Able and willing to complete the informed consent/assent process
* Able and willing to complete the Assessment of Understanding and to verbalize understanding of all questions answered incorrectly prior to signing consent/assent
* Willing to donate blood and urine to be stored and used for future research
* In good general health without clinically significant medical history
* Physical examination and laboratory results without clinically significant findings within the 56 days prior to randomization
* Weight >30 kilograms (kg)
* Agree not to receive any licensed or investigational flavivirus vaccines through 4 weeks after last product administration

Laboratory Criteria within 56 days prior to randomization:

* Hemoglobin within site institutional normal limits
* Absolute neutrophil count (ANC) within site institutional normal limits
* Total lymphocyte count ≥800 cells/mm^3
* Platelets = 125,000-510,000 cells/mm^3
* Alanine aminotransferase (ALT) ≤1.5 x upper limit of normal (ULN) based on site institutional normal range for respective age group
* Serum creatinine ≤1.2 x ULN based on site institutional normal range for respective age group
* Negative result on a human immunodeficiency virus (HIV) test that meets local standards for identification of HIV infection

Criteria applicable to women and adolescents of childbearing potential:

* Negative result on a human chorionic gonadotropin pregnancy test (urine or serum) on day of randomization before receiving study product
* Agree to use effective means of birth control from at least 21 days before randomization through 12 weeks after the last product administration

Criteria applicable to adolescents:

* Capability of the parent/guardian of the minor to understand and comply with planned study procedures
* Capability of the minor and their parent/guardian to provide informed consent/assent

Exclusion Criteria:

Criteria applicable to women and adolescents of childbearing potential:

• Breast-feeding or planning to become pregnant while participating through 12 weeks after the last product administration

Participant has received any of the following:

* More than 10 days of systemic immunosuppressive medications or cytotoxic medications within the 4 weeks prior to randomization
* Any systemic immunosuppressive medications or cytotoxic medications within the 14 days prior to randomization
* Blood products within 16 weeks prior to randomization
* Immunoglobulin within 8 weeks prior to randomization
* Investigational research agents within 4 weeks prior to randomization or planning to receive investigational products while on the study
* Any vaccination within 2 weeks prior to randomization
* Any live attenuated vaccination within 4 weeks prior to randomization
* Current anti-tuberculosis (TB) prophylaxis or therapy

Participant has any of the following:

* Confirmed history of ZIKV infection (as reported by participant)
* Serious reactions to vaccines
* Chronic angioedema or chronic urticaria
* Asthma that is not well-controlled
* Diabetes mellitus (type I or II)
* Clinically significant autoimmune disease or immunodeficiency
* Hypertension that is not well-controlled
* Bleeding disorder diagnosed by a doctor (e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions)
* Significant bruising or bleeding difficulties with IM injections or blood draws
* Malignancy that is active or history of a malignancy that is likely to recur during the period of the study
* Seizure or treatment for a seizure disorder within the last 3 years
* Asplenia, functional asplenia or any condition resulting in the absence or removal of the spleen
* History of Guillain-Barré Syndrome
* Psychiatric condition that may preclude compliance with the protocol; past or present psychoses; or a history of suicide plan or attempt within 5 years prior to randomization
* Any medical psychiatric, or social condition that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a participant's ability to give informed consent

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2428 (Actual)
Dates: Start 2017-03-29 (Actual); Primary Completion 2019-10-04 (Actual); Study Completion 2019-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Ledgerwood, DO, Study Chair — VRC, NIAID, NIH
Locations (17):
- United States (3):
  - QPS-Miami Research Associates, Miami, Florida
  - Doctors Hospital at Renaissance, Edinburg, Texas
  - Baylor College of Medicine, Houston, Texas
- Brazil (2):
  - Hospital Das Clinicas Da Universidade Federal de Minas Gerais, Belo Horizonte, Minas Gerais
  - Centro de Pesquisas Clínicas Do Instituto Central Do Hospital Das Clínicas Da FMUSP, São Paulo, São Paulo
- Colombia (2):
  - Clinica de la Costa Ltda, Barranquilla, Atlántico
  - Centro de Atencion y Diagnostico de Enfermedades Infecciosas, Bucaramanga, Santander Department
- CCIM Costa Rican Center Center of Medical Research, Sociedad Anonima, San José, Los Yoses, Costa Rica
- AGA Clinical Centro de Investigaciones, Guayaquil, Guayas, Ecuador
- Hospital Civil Fray Antonio Alcalde, Guadalajara, Jalisco, Mexico
- Instituto Conmemorativo Gorgas, Panama City, San Miguelito Province, Panama
- Peru (2):
  - Asociacion Civil Selva Amazonica, Iquitos, Maynas/Loreto
  - Unidad de Ensayos (UNIDEC) del Policlinico Universidad Nacional Mayor de San Marcos, Lima
- Puerto Rico (4):
  - Ponce Medical School Foundation Inc./CAIMED Center, Ponce
  - Fundación de Investigación de Diego, San Juan
  - San Juan Hospital Research Unit, San Juan
  - Puerto Rico Clinical and Translational Research Consortium, San Juan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ledgerwood JE, Pierson TC, Hubka SA, Desai N, Rucker S, Gordon IJ, Enama ME, Nelson S, Nason M, Gu W, Bundrant N, Koup RA, Bailer RT, Mascola JR, Nabel GJ, Graham BS; VRC 303 Study Team. A West Nile virus DNA vaccine utilizing a modified promoter induces neutralizing antibody in younger and older healthy adults in a phase I clinical trial. J Infect Dis. 2011 May 15;203(10):1396-404. doi: 10.1093/infdis/jir054. Epub 2011 Mar 11. PMID 21398392
- [Background] Martin JE, Pierson TC, Hubka S, Rucker S, Gordon IJ, Enama ME, Andrews CA, Xu Q, Davis BS, Nason M, Fay M, Koup RA, Roederer M, Bailer RT, Gomez PL, Mascola JR, Chang GJ, Nabel GJ, Graham BS. A West Nile virus DNA vaccine induces neutralizing antibody in healthy adults during a phase 1 clinical trial. J Infect Dis. 2007 Dec 15;196(12):1732-40. doi: 10.1086/523650. PMID 18190252
- [Background] Dowd KA, Ko SY, Morabito KM, Yang ES, Pelc RS, DeMaso CR, Castilho LR, Abbink P, Boyd M, Nityanandam R, Gordon DN, Gallagher JR, Chen X, Todd JP, Tsybovsky Y, Harris A, Huang YS, Higgs S, Vanlandingham DL, Andersen H, Lewis MG, De La Barrera R, Eckels KH, Jarman RG, Nason MC, Barouch DH, Roederer M, Kong WP, Mascola JR, Pierson TC, Graham BS. Rapid development of a DNA vaccine for Zika virus. Science. 2016 Oct 14;354(6309):237-240. doi: 10.1126/science.aai9137. Epub 2016 Sep 22. PMID 27708058
- [Background] Gaudinski MR, Houser KV, Morabito KM, Hu Z, Yamshchikov G, Rothwell RS, Berkowitz N, Mendoza F, Saunders JG, Novik L, Hendel CS, Holman LA, Gordon IJ, Cox JH, Edupuganti S, McArthur MA, Rouphael NG, Lyke KE, Cummings GE, Sitar S, Bailer RT, Foreman BM, Burgomaster K, Pelc RS, Gordon DN, DeMaso CR, Dowd KA, Laurencot C, Schwartz RM, Mascola JR, Graham BS, Pierson TC, Ledgerwood JE, Chen GL; VRC 319; VRC 320 study teams. Safety, tolerability, and immunogenicity of two Zika virus DNA vaccine candidates in healthy adults: randomised, open-label, phase 1 clinical trials. Lancet. 2018 Feb 10;391(10120):552-562. doi: 10.1016/S0140-6736(17)33105-7. Epub 2017 Dec 5. PMID 29217376

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Part A targeted healthy adults only. Part B included adolescents in the study population. Part B sites had the option to enroll adolescents and adults, or choose to enroll only adults. The study was conducted at sites located in areas of confirmed or projected active transmission of Zika virus (ZIKV) infection.
Period: Overall Study
Arm/Group | Part A, Group 1: VRC-ZKADNA090-00-VP (4 mg), 2 Injections | Part A, Group 2: VRC-ZKADNA090-00-VP (4 mg), 4 Injections | Part A, Group 3: VRC-ZKADNA090-00-VP (8 mg), 4 Injections | Part B, Group 4: VRC-ZKADNA090-00-VP (4 mg), 2 Injections | Part B, Group 5: Placebo (VRC-PBSPLA043-00-VP), 2 Injections
Started | 30 | 30 | 30 | 1170 | 1168
Received First Product Administration | 30 | 30 | 30 | 1162 | 1161
Received Second Product Administration | 30 | 29 | 29 | 1126 | 1127
Received Third Product Administration | 29 | 27 | 28 | 1107 | 1107
Completed | 24 | 30 | 28 | 1037 | 1045
Not Completed | 6 | 0 | 2 | 133 | 123
Not completed — Death | 1 | 0 | 0 | 1 | 0
Not completed — Enrolled but did not receive product | 0 | 0 | 0 | 8 | 7
Not completed — Lost to Follow-up | 0 | 0 | 0 | 53 | 45
Not completed — Investigator Decision | 0 | 0 | 0 | 5 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 24 | 24
Not completed — Moved from area | 5 | 0 | 2 | 42 | 43
Not completed — Illness/Injury unrelated to product | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Population includes all randomized subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A, Group 1: VRC-ZKADNA090-00-VP (4 mg), 2 Injections | Part A, Group 2: VRC-ZKADNA090-00-VP (4 mg), 4 Injections | Part A, Group 3: VRC-ZKADNA090-00-VP (8 mg), 4 Injections | Part B, Group 4: VRC-ZKADNA090-00-VP (4 mg), 2 Injections | Part B, Group 5: Placebo (VRC-PBSPLA043-00-VP), 2 Injections | Total
Number analyzed (Participants) | 30 | 30 | 30 | 1170 | 1168 | 2428
Age, Customized [Count of Participants; unit: Participants]
  15-17 years | NA — Part A enrolled healthy adults only and did not include adolescents. | NA — Part A enrolled healthy adults only and did not include adolescents. | NA — Part A enrolled healthy adults only and did not include adolescents. | 17 | 17 | NA — Total not calculated because data are not available (NA) in one or more arms.
  18-20 years | 0 | 0 | 2 | 223 | 222 | 447
  21-30 years | 19 | 24 | 22 | 740 | 734 | 1539
  31-35 years | 11 | 6 | 6 | 190 | 195 | 408
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 22 | 13 | 595 | 601 | 1245
  Male | 16 | 8 | 17 | 575 | 567 | 1183
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 18 | 17 | 1150 | 1139 | 2339
  Not Hispanic or Latino | 15 | 12 | 13 | 17 | 25 | 82
  Unknown or Not Reported | 0 | 0 | 0 | 3 | 4 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 7 | 5 | 6 | 6 | 30
  Asian | 4 | 2 | 1 | 2 | 3 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 0 | 1
  Black or African American | 4 | 2 | 2 | 52 | 41 | 101
  White | 13 | 15 | 17 | 270 | 278 | 593
  More than one race | 3 | 4 | 5 | 834 | 837 | 1683
  Unknown or Not Reported | 0 | 0 | 0 | 5 | 3 | 8
Weight [Mean (Standard Deviation); unit: kilograms] | 86.31 (28.22) | 79.57 (19.84) | 78.55 (23.82) | 70.80 (16.94) | 70.05 (17.49) | 70.84 (17.65)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Local Reactogenicity Signs and Symptoms for 7 Days After Each Product Administration (Part A and Part B)
Description: Participants recorded the occurrence of solicited symptoms on a diary card for 7 days after each study product administration and reviewed the diary card with clinic staff at a follow up visit. Participants were counted once for each symptom at the worst severity if they indicated experiencing the symptom more than one time at any severity during the reporting period. The number reported for "Any Local Symptom" is the number of participants reporting any local symptom at the worst severity. Reactogenicity grading (Mild, Moderate, Severe) was done using the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials (FDA Guidance - September 2007).
Time Frame: 7 days after each product administration
Population: All randomized participants in the study who received at least one study product administration with available data for at least one post-administration assessment for the symptom being summarized.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: VRC-ZKADNA090-00-VP (4 mg), 2 Injections | Part A, Group 2: VRC-ZKADNA090-00-VP (4 mg), 4 Injections | Part A, Group 3: VRC-ZKADNA090-00-VP (8 mg), 4 Injections | Part B, Group 4: VRC-ZKADNA090-00-VP (4 mg), 2 Injections | Part B, Group 5: Placebo (VRC-PBSPLA043-00-VP), 2 Injections
Number analyzed (Participants) | 30 | 30 | 30 | 1153 | 1148
Participants
  Pain/Tenderness: None | 5 | 2 | 2 | 291 | 566
  Pain/Tenderness: Mild | 21 | 21 | 14 | 600 | 482
  Pain/Tenderness: Moderate | 4 | 7 | 14 | 257 | 96
  Pain/Tenderness: Severe | 0 | 0 | 0 | 5 | 4
  Swelling: None | 26 | 25 | 23 | 1059 | 1124
  Swelling: Mild | 4 | 5 | 6 | 82 | 22
  Swelling: Moderate | 0 | 0 | 1 | 12 | 2
  Swelling: Severe | 0 | 0 | 0 | 0 | 0
  Redness: None | 24 | 26 | 23 | 1037 | 1085
  Redness: Mild | 5 | 3 | 7 | 103 | 52
  Redness: Moderate | 1 | 1 | 0 | 13 | 11
  Redness: Severe | 0 | 0 | 0 | 0 | 0
  Any Local Symptom: None | 5 | 2 | 2 | 282 | 552
  Any Local Symptom: Mild | 21 | 20 | 14 | 598 | 485
  Any Local Symptom: Moderate | 4 | 8 | 14 | 268 | 107
  Any Local Symptom: Severe | 0 | 0 | 0 | 5 | 4

2. Primary Outcome: Number of Participants Reporting Systemic Reactogenicity Signs and Symptoms for 7 Days After Each Product Administration (Part A and Part B)
Description: Participants recorded the occurrence of solicited symptoms on a diary card for 7 days after each study product administration and reviewed the diary card with clinic staff at a follow up visit. Participants were counted once for each symptom at the worst severity if they indicated experiencing the symptom more than once at any severity during the reporting period. The number reported for "Any Systemic Symptom" is the number of participants reporting any systemic symptom at the worst severity. Reactogenicity grading (Mild, Moderate, Severe) was done using the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials (FDA Guidance - September 2007).
Time Frame: 7 days after each product administration
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: VRC-ZKADNA090-00-VP (4 mg), 2 Injections | Part A, Group 2: VRC-ZKADNA090-00-VP (4 mg), 4 Injections | Part A, Group 3: VRC-ZKADNA090-00-VP (8 mg), 4 Injections | Part B, Group 4: VRC-ZKADNA090-00-VP (4 mg), 2 Injections | Part B, Group 5: Placebo (VRC-PBSPLA043-00-VP), 2 Injections
Number analyzed (Participants) | 30 | 30 | 30 | 1153 | 1148
Participants
  Malaise: None | 20 | 20 | 17 | 748 | 772
  Malaise: Mild | 8 | 6 | 12 | 306 | 286
  Malaise: Moderate | 2 | 3 | 1 | 97 | 86
  Malaise: Severe | 0 | 1 | 0 | 2 | 4
  Myalgia: None | 26 | 22 | 20 | 793 | 842
  Myalgia: Mild | 3 | 6 | 8 | 270 | 227
  Myalgia: Moderate | 1 | 2 | 2 | 86 | 77
  Myalgia: Severe | 0 | 0 | 0 | 4 | 2
  Headache: None | 20 | 15 | 17 | 696 | 713
  Headache: Mild | 8 | 13 | 13 | 320 | 298
  Headache: Moderate | 2 | 2 | 0 | 131 | 124
  Headache: Severe | 0 | 0 | 0 | 6 | 13
  Chills: None | 27 | 25 | 29 | 1015 | 1029
  Chills: Mild | 3 | 4 | 1 | 109 | 84
  Chills: Moderate | 0 | 1 | 0 | 28 | 33
  Chills: Severe | 0 | 0 | 0 | 1 | 2
  Nausea: None | 26 | 26 | 26 | 971 | 991
  Nausea: Mild | 2 | 3 | 4 | 136 | 118
  Nausea: Moderate | 2 | 1 | 0 | 44 | 34
  Nausea: Severe | 0 | 0 | 0 | 2 | 5
  Joint Pain: None | 26 | 23 | 28 | 964 | 982
  Joint Pain: Mild | 3 | 5 | 2 | 149 | 121
  Joint Pain: Moderate | 1 | 2 | 0 | 36 | 41
  Joint Pain: Severe | 0 | 0 | 0 | 4 | 4
  Fever: None | 30 | 30 | 29 | 1090 | 1082
  Fever: Mild | 0 | 0 | 1 | 37 | 31
  Fever: Moderate | 0 | 0 | 0 | 22 | 24
  Fever: Severe | 0 | 0 | 0 | 4 | 11
  Any Systemic Symptom: None | 16 | 13 | 8 | 508 | 542
  Any Systemic Symptom: Mild | 10 | 12 | 19 | 421 | 394
  Any Systemic Symptom: Moderate | 4 | 4 | 3 | 210 | 190
  Any Systemic Symptom: Severe | 0 | 1 | 0 | 14 | 22

3. Primary Outcome: Number of Participants With Abnormal Laboratory Measures of Safety (Part A)
Description: Any abnormal laboratory results recorded as unsolicited AEs are summarized. Safety laboratory parameters included: alanine aminotransferase (ALT), white blood cells (WBC), red blood cells (RBC), hemoglobin, hematocrit, mean corpuscular volume (MCV), platelets, neutrophils, lymphocytes, monocytes, eosinophils, and basophils. Laboratory safety evaluations were scheduled at baseline and weeks 4, 6, 8, 10, 12, and 16. Institutional laboratory normals as well as the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventative Vaccine Clinical Trials FDA Guidance, September 2007 were used.
Time Frame: Day 0 after first product administration through Day 112
Population: All randomized participants in the study who received at least one study product administration, and had at least one post-administration safety assessment, analyzed according to the study product received.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: VRC-ZKADNA090-00-VP (4 mg), 2 Injections | Part A, Group 2: VRC-ZKADNA090-00-VP (4 mg), 4 Injections | Part A, Group 3: VRC-ZKADNA090-00-VP (8 mg), 4 Injections
Number analyzed (Participants) | 30 | 30 | 30
Participants
  ALT | 3 | 1 | 3
  WBC | 2 | 1 | 3
  Hemoglobin | 2 | 2 | 2
  Platelets | 0 | 1 | 1
  Neutrophil | 0 | 1 | 2
  Lymphocyte | 1 | 0 | 1
  Eosinophil | 1 | 0 | 1

4. Primary Outcome: Number of Participants With Abnormal Laboratory Measures of Safety (Part B)
Description: Any abnormal laboratory results recorded as unsolicited AEs are summarized. Safety laboratory parameters included: alanine aminotransferase (ALT), white blood cells (WBC), red blood cells (RBC), hemoglobin, hematocrit, mean corpuscular volume (MCV), platelets, neutrophils, lymphocytes, monocytes, eosinophils, and basophils. Laboratory safety evaluations were scheduled at baseline and weeks 4, 8, 16, and 44. Institutional laboratory normals as well as the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventative Vaccine Clinical Trials FDA Guidance, September 2007 were used.
Time Frame: Day 0 after first product administration through Day 308
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Part B, Group 4: VRC-ZKADNA090-00-VP (4 mg), 2 Injections | Part B, Group 5: Placebo (VRC-PBSPLA043-00-VP), 2 Injections
Number analyzed (Participants) | 1162 | 1161
Participants
  ALT | 87 | 90
  WBC | 53 | 70
  Hemoglobin | 49 | 53
  Platelets | 7 | 3
  Neutrophil | 19 | 15
  Lymphocyte | 13 | 6
  Eosinophil | 72 | 68

5. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs) Following Product Administration (Part A)
Description: Any SAEs recorded from receipt of first study product administration through the last expected study visit at Day 224 are summarized. The relationship between a SAE and the study product was assessed by the investigator on the basis of his or her clinical judgment and the definitions outlined in the protocol.
Time Frame: Day 0 through Day 224
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: VRC-ZKADNA090-00-VP (4 mg), 2 Injections | Part A, Group 2: VRC-ZKADNA090-00-VP (4 mg), 4 Injections | Part A, Group 3: VRC-ZKADNA090-00-VP (8 mg), 4 Injections
Number analyzed (Participants) | 30 | 30 | 30
Participants
  Related to Study Product | 0 | 0 | 0
  Unrelated to Study Product | 1 | 2 | 0

6. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs) Following Product Administration (Part B)
Description: Any SAEs recorded from receipt of first study product administration through the last expected study visit at Day 672 are summarized. The relationship between a SAE and the study product was assessed by the investigator on the basis of his or her clinical judgment and the definitions outlined in the protocol.
Time Frame: Day 0 through Day 672
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Part B, Group 4: VRC-ZKADNA090-00-VP (4 mg), 2 Injections | Part B, Group 5: Placebo (VRC-PBSPLA043-00-VP), 2 Injections
Number analyzed (Participants) | 1162 | 1161
Participants
  Related to Study Product | 0 | 0
  Unrelated to Study Product | 17 | 18

7. Primary Outcome: Number of Participants With New Chronic Medical Conditions Following Product Administration (Part A)
Description: New onset chronic medical conditions were reported from receipt of first study product administration through the last expected study visit at Day 224.The relationship between a chronic medical condition and the study product was assessed by the investigator on the basis of his or her clinical judgment and the definitions outlined in the protocol.
Time Frame: Day 0 through Day 224
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: VRC-ZKADNA090-00-VP (4 mg), 2 Injections | Part A, Group 2: VRC-ZKADNA090-00-VP (4 mg), 4 Injections | Part A, Group 3: VRC-ZKADNA090-00-VP (8 mg), 4 Injections
Number analyzed (Participants) | 30 | 30 | 30
Participants
  Related to Study Product | 0 | 0 | 0
  Unrelated to Study Product | 0 | 1 | 0

8. Primary Outcome: Number of Participants With New Chronic Medical Conditions Following Product Administration (Part B)
Description: New onset chronic medical conditions were reported from receipt of first study product administration through the last expected study visit at Day 672.The relationship between a chronic medical condition and the study product was assessed by the investigator on the basis of his or her clinical judgment and the definitions outlined in the protocol.
Time Frame: Day 0 through Day 672
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Part B, Group 4: VRC-ZKADNA090-00-VP (4 mg), 2 Injections | Part B, Group 5: Placebo (VRC-PBSPLA043-00-VP), 2 Injections
Number analyzed (Participants) | 1162 | 1161
Participants
  Related to Study Product | 0 | 0
  Unrelated to Study Product | 15 | 9

9. Primary Outcome: Number of Participants With One or More Unsolicited Non-Serious Adverse Events (AEs) Following Product Administration (Part A and Part B)
Description: Unsolicited AEs and attribution assessments were recorded in the study database from receipt of the first study product administration through the one month visit that followed the last study product administration (Visit 05), 84 days for both Parts A and B for participants who received all three study product administrations. If a participant received the first and second product administrations but not the third, then the time frame was through 56 days (Visit 04). If a participant only received the first product administration but not the second or third, then the time frame was through 28 days (Visit 03). The relationship between an AE and the study product was assessed by the investigator on the basis of his or her clinical judgment and the definitions outlined in the protocol. A participant with multiple experiences of the same event is counted once using the event of worst severity.
Time Frame: Day 0 through the one month visit that follows the last product administration (Visit 05), 84 days for both Parts A and B
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: VRC-ZKADNA090-00-VP (4 mg), 2 Injections | Part A, Group 2: VRC-ZKADNA090-00-VP (4 mg), 4 Injections | Part A, Group 3: VRC-ZKADNA090-00-VP (8 mg), 4 Injections | Part B, Group 4: VRC-ZKADNA090-00-VP (4 mg), 2 Injections | Part B, Group 5: Placebo (VRC-PBSPLA043-00-VP), 2 Injections
Number analyzed (Participants) | 30 | 30 | 30 | 1162 | 1161
Participants
  Related to Study Product | 4 | 5 | 6 | 77 | 58
  Unrelated to Study Product | 18 | 14 | 20 | 500 | 530

10. Primary Outcome: Number of Participants With Virologically Confirmed Cases of ZIKV (Part B Only)
Description: Virologically confirmed Zika infection, irrespective of symptoms, by polymerase chain reaction (PCR) in blood or in urine were recorded from receipt of first study product administration through the last expected study visit.
Time Frame: Day 0 through Day 672
Population: All randomized participants in the study, analyzed according to the randomized study product. One placebo participant, who had a virologically confirmed case of ZIKV from a sample collected prior to first product administration, is not counted as a virologically confirmed case.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B, Group 4: VRC-ZKADNA090-00-VP (4 mg), 2 Injections | Part B, Group 5: Placebo (VRC-PBSPLA043-00-VP), 2 Injections
Number analyzed (Participants) | 1170 | 1168
Participants | 1 | 2

11. Secondary Outcome: Zika Antigen-specific Neutralizing Antibody Geometric Mean Titer (GMT) - (Part A)
Description: Antibody response as measured by ZIKV neutralization antibody (NAb) assay. Neutralizing activity is reported as the dilution of sera required to neutralize eighty percent of infection events (EC80).
Time Frame: Day 0 to 28 days after the third product administration
Population: All randomized participants, analyzed according to the randomized study product. All participants with samples at the protocol-defined immunogenicity timepoint were analyzed. The two subjects missing from Group 1 missed their Day 28 visit and thus there was no sample to analyze.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Part A, Group 1: VRC-ZKADNA090-00-VP (4 mg), 2 Injections | Part A, Group 2: VRC-ZKADNA090-00-VP (4 mg), 4 Injections | Part A, Group 3: VRC-ZKADNA090-00-VP (8 mg), 4 Injections
Number analyzed (Participants) | 28 | 30 | 30
titer
  Day 0 (Baseline, Pre-administration) | 22.288 [15.056 to 32.994] | 34.836 [19.903 to 60.973] | 22.25 [14.948 to 33.121]
  Day 28 After the Third Product Administration | 77.468 [46.696 to 128.516] | 187.629 [117.826 to 298.785] | 130.497 [90.082 to 189.043]

12. Secondary Outcome: Number of Participants With Positive Response to Zika Antigen-specific Neutralizing Antibody (Part A)
Description: A participant was a responder or met the threshold of a positive response if the post vaccination anti-ZIKV antibody titer was 30 or greater.
Time Frame: Day 0 to 28 days after the third product administration
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: VRC-ZKADNA090-00-VP (4 mg), 2 Injections | Part A, Group 2: VRC-ZKADNA090-00-VP (4 mg), 4 Injections | Part A, Group 3: VRC-ZKADNA090-00-VP (8 mg), 4 Injections
Number analyzed (Participants) | 28 | 30 | 30
Participants
  Day 0 (Baseline, Pre-administration) | 5 | 8 | 4
  Day 28 After the Third Product Administration | 20 | 27 | 29

13. Secondary Outcome: Number of Participants With Subclinical Cases of ZIKV (Part B Only)
Description: Virologically confirmed cases of Zika infection without clinical signs or symptoms were recorded from receipt of first study product administration through the last expected study visit by PCR virus detection in blood of participants at regularly defined intervals. Subclinical cases of ZIKV infection were identified by retrospective PCR.
Time Frame: Day 0 through Day 672
Population: All randomized participants in the study, analyzed according to the randomized study product. One placebo participant had a subclinical case of ZIKV from a sample collected prior to first product administration. Two placebo participants had subclinical cases of ZIKV but also reported symptomatic ZIKV cases close in time to the positive subclinical result, consistent with a clinical picture of one symptomatic ZIKV infection event for each. These 3 are not counted as subclinical cases.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B, Group 4: VRC-ZKADNA090-00-VP (4 mg), 2 Injections | Part B, Group 5: Placebo (VRC-PBSPLA043-00-VP), 2 Injections
Number analyzed (Participants) | 1170 | 1168
Participants | 1 | 0

14. Secondary Outcome: Zika Antigen-specific Neutralizing Antibody Geometric Mean Titer (GMT) - (Part B)
Description: Antibody response as measured by ZIKV neutralization antibody (NAb) assay. Neutralizing activity is reported as the dilution of sera required to neutralize fifty percent of infection events (EC50).
Time Frame: Day 0 to 28 days after the third product administration
Population: Subset of per protocol population, which included randomly selected study participants who received three administrations within window as assigned by the randomization schedule and did not have any other major protocol deviations prior to their Week 12 visit, was analyzed to meet statistical power.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Part B, Group 4: VRC-ZKADNA090-00-VP (4 mg), 2 Injections | Part B, Group 5: Placebo (VRC-PBSPLA043-00-VP), 2 Injections
Number analyzed (Participants) | 143 | 51
titer
  Day 0 (Baseline, Pre-administration) | 94.7 [68.5 to 131.1] | 205.3 [113.0 to 373.2]
  Day 28 After the Third Product Administration | 567.7 [448.3 to 718.9] | 191.9 [108.1 to 340.8]

15. Secondary Outcome: Number of Participants With Positive Response to Zika Antigen-specific Neutralizing Antibody (Part B)
Description: A participant is a responder or met the threshold of a positive response if the post vaccination anti-ZIKV antibody titer was 30 or greater.
Time Frame: Day 0 to 28 days after the third product administration
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Part B, Group 4: VRC-ZKADNA090-00-VP (4 mg), 2 Injections | Part B, Group 5: Placebo (VRC-PBSPLA043-00-VP), 2 Injections
Number analyzed (Participants) | 143 | 51
Participants
  Day 0 (Baseline, Pre-administration) | 80 | 35
  Day 28 After the Third Product Administration | 139 | 35

ADVERSE EVENTS:
Time Frame: Solicited adverse events (AEs) were reported for 7 days after each study injection. Unsolicited AEs were recorded from receipt of the first study injection through the one month visit that followed the last product administration. At other time periods, only SAEs, new chronic medical conditions and confirmed cases of Dengue (DENV) infection were recorded through the last expected study visit (Part A: Day 224 and Part B: Day 672).
Description: Solicited AEs collected through systematic assessment and unsolicited AEs collected through non-systematic assessment were recorded for subjects who received at least one study injection and provided safety data following the injection, and represent the number and percentage of subjects reporting the event. A subject with multiple experiences of the same event is counted once using the event of worst severity.
Arm/Group | Part A, Group 1: VRC-ZKADNA090-00-VP (4 mg), 2 Injections | Part A, Group 2: VRC-ZKADNA090-00-VP (4 mg), 4 Injections | Part A, Group 3: VRC-ZKADNA090-00-VP (8 mg), 4 Injections | Part B, Group 4: VRC-ZKADNA090-00-VP (4 mg), 2 Injections | Part B, Group 5: Placebo (VRC-PBSPLA043-00-VP), 2 Injections
All-Cause Mortality (participants affected / at risk) | 1/30 | 0/30 | 0/30 | 1/1162 | 0/1161
Serious Adverse Events (participants affected / at risk) | 1/30 | 2/30 | 0/30 | 17/1162 | 18/1161
Other Adverse Events (participants affected / at risk) | 28/30 | 29/30 | 30/30 | 990/1162 | 859/1161
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A, Group 1: VRC-ZKADNA090-00-VP (4 mg), 2 Injections (N=30) | Part A, Group 2: VRC-ZKADNA090-00-VP (4 mg), 4 Injections (N=30) | Part A, Group 3: VRC-ZKADNA090-00-VP (8 mg), 4 Injections (N=30) | Part B, Group 4: VRC-ZKADNA090-00-VP (4 mg), 2 Injections (N=1162) | Part B, Group 5: Placebo (VRC-PBSPLA043-00-VP), 2 Injections (N=1161)
Atrial septal defect (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 — The congenital anomaly/birth defects were in the offspring of the participant.
Congenital hydronephrosis (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 — The congenital anomaly/birth defects were in the offspring of the participant.
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 2 | 4
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Cellulitis orbital (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pelvic inflammatory disease (Infections and infestations) | 0 | 0 | 0 | 2 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Gun shot wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2
Mucinous cystadenocarcinoma ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1
Bipolar disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Conversion disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 2 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A, Group 1: VRC-ZKADNA090-00-VP (4 mg), 2 Injections (N=30) | Part A, Group 2: VRC-ZKADNA090-00-VP (4 mg), 4 Injections (N=30) | Part A, Group 3: VRC-ZKADNA090-00-VP (8 mg), 4 Injections (N=30) | Part B, Group 4: VRC-ZKADNA090-00-VP (4 mg), 2 Injections (N=1162) | Part B, Group 5: Placebo (VRC-PBSPLA043-00-VP), 2 Injections (N=1161)
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 2 | 51 | 56
Leukocytosis (Blood and lymphatic system disorders) | 2 | 1 | 1 | 49 | 67
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 4 | 3
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 2 | 19 | 15
Bradycardia (Cardiac disorders) | 1 | 1 | 2 | 21 | 24
Nausea (Gastrointestinal disorders) | 4 | 4 | 4 | 182 | 157
Administration site erythema (General disorders) | 6 | 4 | 7 | 116 | 63 — Redness
Administration site pain (General disorders) | 25 | 28 | 28 | 862 | 582
Administration site swelling (General disorders) | 4 | 5 | 7 | 94 | 24
Chills (General disorders) | 3 | 5 | 1 | 139 | 119
Injection site bruising (General disorders) | 5 | 10 | 13 | 31 | 26
Injection site pruritus (General disorders) | 1 | 1 | 2 | 12 | 3
Malaise (General disorders) | 10 | 10 | 13 | 405 | 376
Gastroenteritis (Infections and infestations) | 2 | 0 | 1 | 11 | 17
Pharyngitis (Infections and infestations) | 2 | 0 | 0 | 28 | 22
Sinusitis (Infections and infestations) | 0 | 0 | 2 | 3 | 5
Upper respiratory tract infection (Infections and infestations) | 4 | 1 | 5 | 36 | 35
Viral infection (Infections and infestations) | 2 | 1 | 0 | 21 | 26
Alanine aminotransferase increased (Investigations) | 3 | 1 | 3 | 87 | 92
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 7 | 2 | 189 | 167 — Joint Pain
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 8 | 10 | 362 | 306
Headache (Nervous system disorders) | 10 | 14 | 13 | 444 | 432
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 4 | 3
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 2 | 3
Hypertension (Vascular disorders) | 0 | 1 | 3 | 26 | 27
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 72 | 69
Pyrexia (General disorders) | 0 | 0 | 1 | 63 | 66 — Fever (Temperature)
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 72 | 75
Headache (Nervous system disorders) | 0 | 1 | 2 | 21 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-11-11): https://cdn.clinicaltrials.gov/large-docs/70/NCT03110770/Prot_SAP_ICF_000.pdf